CLINICAL TRIAL: NCT05649904
Title: Use of Active Fluid Exchange to Therapeutically Treat Intracranial Bleeding and Infection
Brief Title: AFFECT Study for Patients With Intraventricular Hemorrhage, Subarachnoid Hemorrhage, Subdural Hematoma, and Ventriculitis
Acronym: AFFECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: IRRAS (Industry)
Responsible Party: Principal Investigator, Patrick Youssef, Clinical Assistant Professor of Neurological Surgery, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022H0197
Record Dates: First submitted 2022-10-24; First posted 2022-12-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Intraventricular Hemorrhage; Subarachnoid Hemorrhage; Subdural Hematoma; Ventriculitis
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hematoma, Subdural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IRRAflow with Active Fluid Exchange System (IRRAflow) (Experimental): Subjects may be randomized to receive the IRRAflow with Active Fluid Exchange System (intervention) for intracranial pressure monitoring and for externally draining intracranial fluid as a means of reducing intracranial pressure.
  Interventions: Device: IRRAflow with Active Fluid Exchange System
- External Ventricular Drainage (EVD) (Active Comparator): Subjects may be randomized to receive an External Ventricular Drain (control) for intracranial pressure monitoring and for externally draining intracranial fluid as a means of reducing intracranial pressure.
  Interventions: Device: External Ventricular Drain

INTERVENTIONS:
Device: IRRAflow with Active Fluid Exchange System — IRRAflow® Active Fluid Exchange System is an intracranial drainage system intended for use by professional medical hospital personnel, trained and experienced in neurosurgical medical care.
  The intracranial pressure is kept at a safe level by draining excessive intracranial fluid. The system incorporates an irrigation support mechanism, used to irrigate the system in a controlled, programmed manner to minimize catheter occlusion. Additionally, a manual bolus can be given to facilitate keeping the catheter clear of occlusion or to clear the catheter of occlusion if one is present. This mechanism works by producing a bolus pulse using short periods of high flow (i.e. flow pulses).
  Other Names: IRRAflow
  Arms: IRRAflow with Active Fluid Exchange System (IRRAflow)
Device: External Ventricular Drain — The External Ventricular Drain (EVD) is used standard of care at the study site for ventricular drainage.
  Other Names: EVD
  Arms: External Ventricular Drainage (EVD)

SUMMARY:
The goal of this clinical trial is to evaluate efficacy and safety of evacuation of cerebrospinal fluid, blood, and harmful bacteria from the intraventricular, subdural and subarachnoid spaces by Active Controlled Irrigation and Drainage (IRRAflow) compared to Passive External Ventricular Drainage (EVD).

Subjects with intraventricular hemorrhage, subarachnoid hemorrhage, subdural bleeding, and ventriculitis will be randomized to receive the IRRAflow device or EVD device and followed for one month post-procedure to compare outcomes between the subject groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Need of drainage for one of the following underlying conditions: Intraventricular hemorrhage, intracranial hemorrhage, subarachnoid hemorrhage, chronic subdural hematoma and ventriculitis
3. Indication for active treatment evaluated by treating physician for underlying conditions; Intraventricular hemorrhage, subarachnoid hemorrhage, chronic subdural hematoma and ventriculitis
4. Signed informed consent obtained by subject or Legally Authorized Representative

Exclusion Criteria:

1. Subject has fixed and dilated pupils
2. Pregnant women
3. Presence of Moyamoya
4. History or presence of clotting disorder.
5. Platelet count less than 100,000, INR greater than 1.4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of revision procedures for the IRRAflow and EVD/Drainage catheters | Immediately post-procedure

SECONDARY OUTCOMES:
Time to clearance of blood or bacterial mass as measured by head CT scan | Immediately post-procedure
Rate of catheter-related infection | Immediately post-procedure
Length of ICU stay | Baseline
Rate of shunt dependency | Immediately post-procedure
Indwell time of EVD/Drainage and IRRAflow Catheter | Immediately post-procedure
Functional Status - at inclusion and 30 days | 30 days post subject discharge
  The Modified Rankin Scale will be used to assess functional status. The Modified Rankin Scale ranges from 0 (no disability) to 6 (death).
Mortality rates - intraprocedural and at 30 days | 30 days post subject discharge
Functional Status - at inclusion and 30 days | 30 days post subject discharge
  The Extended Glasgow Coma Scale will be used to assess functional status. Results range from 1 (death) to 8 (upper good recovery).
Functional Status - at inclusion and 30 days | 30 days post subject discharge
  The Barthel Index will be used to assess functional status. Scores for this assessment tool range from 0 - 100, with a higher number indicating a better functional status.
Functional Status - at inclusion and 30 days | 30 days post subject discharge
  The Stroke Impact Scale will be used to assess functional status. Scores for this scale range from 0 - 100, with a higher number indicating a better functional status.
Functional Status - at inclusion and 30 days | 30 days post subject discharge
  The EQ-VAS will be used to assess functional status. Participants rate their health from 0 (worst imaginable health) to 100 (best imaginable health).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Youssef, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No